CLINICAL TRIAL: NCT05158595
Title: Effects of Exergame Balance Training on Dementia-Related Quality of Life and Self-Efficacy in Patients With Mild Cognitive Impairment
Brief Title: Exer-game Balance Training on Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01032/Sehar
Record Dates: First submitted 2021-08-27; First posted 2021-12-15 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low intensity group (Experimental): Will receive wobble board based Exergame balance training, game intensity will be low for this group (Size of goal will be kept large)
  Interventions: Other: Exergaming low intensity group
- moderate intensity group (Experimental): Will receive wobble board based Exergame balance training, game intensity will be low for this group (Size of goal will be kept large)
  Interventions: Other: Exergaming moderate intensity group
- high intensity group (Experimental): Will receive wobble board-based Exergame balance training, game intensity will be high for this group (Size of goal will be kept small).
  Interventions: Other: Exergaming high intensity group
- control group (Active Comparator): Will receive Exer-game balance training with Wii Fit balance games
  Interventions: Other: control group exergaming

INTERVENTIONS:
Other: Exergaming low intensity group — wobble board-based Exergame balance training, the game intensity will be low for this group (Size of goal will be kept small for 3 times a week, 30 minutes per day for 8 weeks.
  Arms: low intensity group
Other: Exergaming moderate intensity group — Wobble board-based Exer- game balance training, the game intensity will be moderate for this group (size of goal will be kept medium).for 3 times a week, 30 minutes per day for 8 weeks.
  Arms: moderate intensity group
Other: Exergaming high intensity group — Wobble board-based Exer- game balance training, the game intensity will be moderate for this group (size of goal will be kept high).for 3 times a week, 30 minutes per day for 8 weeks.
  Arms: high intensity group
Other: control group exergaming — Exer games training with soccer heading and penguin slide games(Wii Fitt balance games) for 3 times a week, 30 minutes per day for 8 weeks.
  Arms: control group

SUMMARY:
Age-related cognitive impairment is a wide phenomenon. Mild cognitive impairment is a transitional stage between Dementia and normal cognition.Mild cognitive impairment (MCI) is a syndrome that has been recognized in older adults and it has become a topic of a major focus on clinical care and research. In people with this condition, there are cognitive deficits and these have adverse effects on activities of daily living . These patients cannot recognize their impairment. Mild cognitive impairment is a risk factor for dementia.

DETAILED DESCRIPTION:
The clinical features of MCI are memory impairment along with language or speech impairments, executive functions, and visuospatial impairments. In regard to clinical features of Mild cognitive impairment (MCI), there are motor problems as patients have difficulty in doing complex motor tasks like doing pegboard assembly and also in fine and gross motor skills performance like they have difficulty in maintaining balance and body weight. Major factors contributing to mild cognitive impairment or major causes are medical conditions like hepatic or renal failure, depression, sleep disturbances, psychological problems,s and medicine side effects. impaired attention and concentration can lead to impaired memory and a decline in cognitive function.

As literature supports the evidence of the effectiveness of Exergaming in adults with neurocognitive disorders.As Exer-gaming training program improved their lower extremity functioning, cognitive function, and reduced depression, neuropsychiatric symptoms too. Recent studies on the treatment of Exergaming and its effect on the quality of life in dementia approach the standing balance Exer-gaming being effective and has increased attention, concentration, memory, and reaction time and has improved physical, cognitive, emotional, social function and quality of life and decreased the level of frailty in dementia patients. Recent literature on Exergaming has successfully improved cognition, balance,gait, and verbal memory in MCI patients and reduced fall risk in older adults of age >55 years

ELIGIBILITY:
Inclusion Criteria:

* Individuals >55 years of age.
* Patients meeting mild cognitive impairment (MCI), The Montreal Cognitive Assessment (MoCA) 20-24.
* clinical dementia rating scale (CDR) ≤ 1.0
* No unstable disease precluding the planned exercise
* Able to see and hear sufficiently to participate in planned physical and computer-based cognitive training

Exclusion Criteria:

* Non-ambulatory or major mobility disorder;
* Other neurological conditions associated with cognitive impairment such as stroke, Parkinson disease, and head injury
* Any clinically significant psychiatric condition, current drug or alcohol abuse, that would interfere with the ability to participate in the study
* Severe visual impairment
* Unwillingness to participate

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
DEMENTIA QUALITY OF LIFE QUESTIONAIRRE (DEMQOL) | week 8
  it has 29 statements with five scales and each scale score is measured by taking mean of the individual items. Every item have a 5-point scale response format on enjoyment (not at all, a lot) and frequency (never, very often).
General Self Efficacy scale | week 8
  This tool tells human behavior and coping outcomes. It's very useful with studying behaviour of people who are living with any illness. This scale have 10-items and possible responses are "not at all ,all true"1=hardly true, 2=moderately true,3= exactly true,4=total score between 10 and 40
2 Minute Walk test (2MWT) | week 8
  is a reliable and valid tool for accessing balance in older adults. Instructions given to the participants are that you have to "walk at your comfortable zone. The assessor will be half a meter behind the participant to ensure his/her safety. No encouragement or feedback is given during the whole test. Two practice trials and one final trial for record are performed. The participants are given at least 10 min rest between trials. The distance covered in the 2 min is recorded as the 2MWT

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Malik, PhD, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussenoeder FS, Conrad I, Roehr S, Fuchs A, Pentzek M, Bickel H, Moesch E, Weyerer S, Werle J, Wiese B, Mamone S, Brettschneider C, Heser K, Kleineidam L, Kaduszkiewicz H, Eisele M, Maier W, Wagner M, Scherer M, Konig HH, Riedel-Heller SG. Mild cognitive impairment and quality of life in the oldest old: a closer look. Qual Life Res. 2020 Jun;29(6):1675-1683. doi: 10.1007/s11136-020-02425-5. Epub 2020 Jan 28. PMID 31993915
- [Background] Griffiths J, Thaikruea L, Wongpakaran N, Munkhetvit P. Prevalence of Mild Cognitive Impairment in Rural Thai Older People, Associated Risk Factors and their Cognitive Characteristics. Dement Geriatr Cogn Dis Extra. 2020 Mar 26;10(1):38-45. doi: 10.1159/000506279. eCollection 2020 Jan-Apr. PMID 32308666
- [Background] Foster NL, Bondi MW, Das R, Foss M, Hershey LA, Koh S, Logan R, Poole C, Shega JW, Sood A, Thothala N, Wicklund M, Yu M, Bennett A, Wang D. Quality improvement in neurology: Mild cognitive impairment quality measurement set. Neurology. 2019 Oct 15;93(16):705-713. doi: 10.1212/WNL.0000000000008259. Epub 2019 Sep 18. No abstract available. PMID 31534026
- [Background] Tangalos EG, Petersen RC. Mild Cognitive Impairment in Geriatrics. Clin Geriatr Med. 2018 Nov;34(4):563-589. doi: 10.1016/j.cger.2018.06.005. Epub 2018 Aug 21. PMID 30336988
- [Background] Mariani E, Monastero R, Mecocci P. Mild cognitive impairment: a systematic review. J Alzheimers Dis. 2007 Aug;12(1):23-35. doi: 10.3233/jad-2007-12104. PMID 17851192
- [Background] Alkhunizan M, Alkhenizan A, Basudan L. Prevalence of Mild Cognitive Impairment and Dementia in Saudi Arabia: A Community-Based Study. Dement Geriatr Cogn Dis Extra. 2018 Mar 20;8(1):98-103. doi: 10.1159/000487231. eCollection 2018 Jan-Apr. PMID 29706986
- [Background] Wada-Isoe K, Uemura Y, Nakashita S, Yamawaki M, Tanaka K, Yamamoto M, Shimokata H, Nakashima K. Prevalence of Dementia and Mild Cognitive Impairment in the Rural Island Town of Ama-cho, Japan. Dement Geriatr Cogn Dis Extra. 2012 Jan;2(1):190-9. doi: 10.1159/000338244. Epub 2012 Apr 24. PMID 22719745
- [Background] Mohan D, Iype T, Varghese S, Usha A, Mohan M. A cross-sectional study to assess prevalence and factors associated with mild cognitive impairment among older adults in an urban area of Kerala, South India. BMJ Open. 2019 Mar 20;9(3):e025473. doi: 10.1136/bmjopen-2018-025473. PMID 30898818
- [Background] Juarez-Cedillo T, Sanchez-Arenas R, Sanchez-Garcia S, Garcia-Pena C, Hsiung GY, Sepehry AA, Beattie BL, Jacova C. Prevalence of mild cognitive impairment and its subtypes in the Mexican population. Dement Geriatr Cogn Disord. 2012;34(5-6):271-81. doi: 10.1159/000345251. Epub 2012 Nov 29. PMID 23207978
- [Background] Vlachos GS, Kosmidis MH, Yannakoulia M, Dardiotis E, Hadjigeorgiou G, Sakka P, Ntanasi E, Stefanis L, Scarmeas N. Prevalence of Mild Cognitive Impairment in the Elderly Population in Greece: Results From the HELIAD Study. Alzheimer Dis Assoc Disord. 2020 Apr-Jun;34(2):156-162. doi: 10.1097/WAD.0000000000000361. PMID 31913961